CLINICAL TRIAL: NCT00965796
Title: Effect of Intraoperative Intravenous Lidocaine on Pain After Hysterectomy
Brief Title: Intraoperative Intravenous Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rioko K Sakata, Universidade Federal de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IO-Lido
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Pain Intensity
Keywords: Intravenous lidocaine; postoperative analgesia
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine, pain intensity and Saline (Experimental): (2 mg/kg/h) and patients of group 2 (n = 20) received 0.9% saline infusion throughout the surgical procedure
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2 mg/kg/h- during surgical procedure Saline
  Other Names: Intravenous lidocaine

SUMMARY:
The objective of the present study was to evaluate the effect of intraoperative intravenous lidocaine on postoperative pain after hysterectomy.

DETAILED DESCRIPTION:
Study design A prospective, randomized, double-blind study was conducted according to ethical guidelines for research involving humans. The study was approved by the Ethics Committee of the institution and all patients signed a free informed consent form. The patients were randomly allocated to two groups consisting of the same number of subjects by drawing lots.

One physician prepared the solutions and handed them over to the anesthetist who was unaware of the content of the solutions. The volume of the solutions was the same. The researcher was unaware to which group the patient belonged until the end of the study.

Exclusion criteria Excluded from the study were patients with cardiac arrhythmia; myocardiopathy; altered cardiac conduction; psychiatric, hepatic or respiratory disease; and patients receiving any type of analgesic during the week before surgery.

Patients Forty women (ASA 1 or 2) aged 18 to 60 years undergoing hysterectomy were studied.

Treatment Patients of group 1 (n = 20) received lidocaine (2 mg/kg/h) and patients of group 2 (n = 20) received 0.9% saline infusion throughout the surgical procedure.

Anesthesia Oral midazolam (15 mg) was administered one hour before anesthesia as pre-anesthetic medication. Anesthesia was induced with 5 µg/kg fentanyl and 2 mg/kg propofol. Neuromuscular block was maintained with atracurium. Anesthesia was maintained with O2/isoflurane.

Patient assessment The supplemental morphine doses necessary during the first 24 h and the time to first analgesic request were recorded. Pain intensity was evaluated at rest on a numerical scale ranging from 0 to 10 (0 = no pain and 10 = most intense pain possible) at the following times: T0 (immediately after arousal), and 6, 12, 18 and 24 h after arousal. Side effects were recorded.

Statistical analysis The results were analyzed statistically with the Instat Graph program using parametric and nonparametric tests, depending on the nature of the variables studied. Measures of central tendency (means) and dispersion (standard deviation) were used. The level of significance was set at < 0.05. The following tests were used: Mann-Whitney test for age, body mass index, duration of anesthesia and surgery, time to first analgesic supplementation, total amount of morphine, pain intensity, and isoflurane consumed; Student t-test for weight and height; and Friedman test for pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2, aged 18 to 60 years undergoing hysterectomy

Exclusion Criteria:

* Cardiac arrhythmia; myocardiopathy
* Altered cardiac conduction
* Psychiatric, hepatic or respiratory disease
* Patients receiving any type of analgesic during the week before surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain | 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (2):
- Brazil (2):
  - Rioko K Sakata- Universidade Federal de São Paulo, São Paulo, Rua Botucatu-593
  - Universidade Federal de São Paulo, São Paulo, São Paulo